CLINICAL TRIAL: NCT00971386
Title: Short Term Hemodynamic Effects of Controlled Slow Breathing With Biofeedback in Patients With Heart Failure: Normal Healthy Subjects vs. Chronic Ambulatory Heart Failure Patients vs Acute Heart Failure
Brief Title: Short Term Hemodynamic Effects of Controlled Slow Breathing With Biofeedback in Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Darshak H. Karia, MD. Director, Heart Failure Services, Albert Einstein Heart and Vascular, Albert Einstein Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HN 4025
Record Dates: First submitted 2009-08-05; First posted 2009-09-03 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal Healthy Subjects (Other): Normal healthy subjects without history, signs-symptoms or diagnosis of heart failure
  Interventions: Behavioral: Slow breathing
- Chronic Ambulatory Heart Failure (Other): Diagnosis of Chronic Heart Failure and currently on optimal medical therapy
  Interventions: Behavioral: Slow breathing
- Acute Heart Failure (Other): Patients admitted to the hospital with acute congestive heart failure.
  Interventions: Behavioral: Slow breathing

INTERVENTIONS:
Behavioral: Slow breathing — The subjects will be given instructions in slow breathing at a rate of 6 to 10 breaths per minute and asked to practice it for some time. Hemodynamic measurements would be repeated before, during and after the trial of slow breathing. A Noninvasive Cardiac Output Monitor will be used. It uses a technology called impedance to measure cardiac output and other hemodynamic parameters by the passage of electric currents through the thorax. This device uses four electrode stickers applied to the thorax and the neck.

SUMMARY:
Heart failure is associated with faster breathing, which has a negative impact on the functioning of the heart. This leads to fatigue, shortness of breath, and exercise intolerance. It has been shown that when slow breathing technique was taught to patients with heart failure, they had a reduction in their sensation of shortness of breath and an improvement in their exercise performance.

The study will compare the short-term effects of controlled slow breathing with biofeedback in normal healthy subjects, acute heart failure, and chronic stable heart failure. The purpose is to see if there is any change in the objective measurements of heart function while breathing at normal rates compared to a controlled slower rate.

DETAILED DESCRIPTION:
Heart Failure (HF) is a growing and challenging public health concern in the United States. Current data suggest that there are about 5 million heart failure patients in this country with an additional 550,000 patients being diagnosed with this syndrome each year for the first time. Despite the significant advances in the management strategy of heart failure patients in the last 1-2 decades, there are about 1 million hospital admissions each year for Acute Decompensated Heart Failure (ADHF), almost double the number seen 15 years ago. The readmission rate for these patients at 6-month following discharge approaches about 50% with estimated 5-year mortality of 50%. Approximately, $23 billion are spent for the inpatient management of HF patients with another $40 billion for outpatient care. This prevailing situation mandates further exploration of novel therapeutic targets to treat this complex disease.

Chronic HF is accompanied by a sustained elevation in sympathetic nervous system activity, which is thought to be an important component in the pathophysiology and progression of the disease. HF patients also show abnormal breathing pattern with an increased respiratory rate and a lower tidal volume. Faster respiratory rate is associated with higher levels of sympathetic activity and potentiation of the chemoreflex response to hypoxia and hypercapnia. The relationship between sympathetic activity and spontaneous breathing rate is independent of age, body mass index, physical activity levels, percentage of body fat, or blood pressure. The arterial baroreflex sensitivity is also reduced in patients with heart failure. All these factors contribute to the distressing symptoms of fatigue, dyspnea and exercise intolerance in these patients.

Yoga trainees learn to breathe slowly, at a rate of about six breaths per minute, mobilizing in sequence the diaphragm and the upper and the lower chest. A handful of studies in normal subjects undergoing intensive training in yogic breathing techniques have demonstrated a marked improvement in cardiac hemodynamic parameters (cardiac output, cardiac index, stroke volume etc.), but such studies have not been conducted in patients with heart failure.

The purpose of our study is to evaluate the changes in cardiac hemodynamic parameters (cardiac output, cardiac index and thoracic fluid content) in patients with acute heart failure, chronic ambulatory heart failure and normal healthy subjects after a trial of controlled slow breathing. Subjects would undergo non-invasive measurement of cardiac hemodynamics while spontaneously breathing. They would then be given instructions in slow breathing at a rate of 6 to 10 breaths per minute and asked to practice it for some time using heart rate variability as biofeedback mechanism. Hemodynamic measurements would be repeated during and after the trial of slow breathing. The difference between these measurements would then be statistically analyzed. We hypothesize that even a short trial of controlled slow breathing using a biofeedback mechanism in patients with HF would produce significant favorable improvement in cardiac hemodynamics.

ELIGIBILITY:
Inclusion Criteria: NORMAL SUBJECTS

1. Normal subject without history, signs-symptoms or diagnosis of heart failure
2. Age over 18 and willing and able to provide informed consent.

Exclusion Criteria: NORMAL SUBJECTS

1. Known allergy to electrode gel and medical adhesive used on electrocardiographic electrodes.
2. Pregnancy (as any effect of this device use on pregnancy is not known).
3. Patient belonging to a vulnerable population such as institutionalized persons, prisoners and persons with decisional incapacity or dementia.
4. Presence of severe aortic regurgitation.
5. Second degree Mobitz type II or third degree heart block, unless treated with a cardiac pacemaker.
6. Implantation of a left ventricular assists device, hemodynamic monitor, activated minute ventilation pacemaker, or biventricular pacemaker (Cardiac Resynchronization Therapy) with the V-to-V interval set at more than 5 milliseconds offset.
7. Implantation of a cardiac resynchronization device within the last 30 days.

Inclusion Criteria: CHRONIC AMBULATORY HEART FAILURE

1. Patients over the age of 18 and able to give consent
2. Ability to understand and willing to sign informed consent
3. Diagnosis of Chronic Heart Failure and currently on optimal medical therapy

Exclusion Criteria: CHRONIC AMBULATORY HEART FAILURE

1. NYHA class III/ IV heart failure symptoms despite treatment with diuretics.
2. Co-existent pulmonary disease such as asthma/ COPD/ interstitial lung disease.
3. Known allergy to electrode gel and medical adhesive used on electrocardiographic electrodes.
4. Pregnancy (as any effect of this device use on pregnancy is not known).
5. Patient belonging to a vulnerable population such as institutionalized persons, prisoners and persons with decisional incapacity or dementia.
6. Presence of severe aortic regurgitation.
7. Second degree Mobitz type II or third degree heart block, unless treated with a cardiac pacemaker.
8. Implantation of a left ventricular assists device, hemodynamic monitor, activated minute ventilation pacemaker, or biventricular pacemaker (Cardiac Resynchronization Therapy) with the V-to-V interval set at more than 5 milliseconds offset.
9. Implantation of a cardiac resynchronization device within the last 30 days.

Inclusion Criteria: ACUTE HEART FAILURE

1. Patients over the age of 18 willing to and able to provide informed consent.
2. Patients admitted to the hospital with acute congestive heart failure (evidenced by pulmonary edema by CXR, BNP> 500 pg/ml, jugular venous distension (JVD), crackles/ rales, dependent edema) who have been stabilized with medical therapy with evidence of euvolemia by at least two of the following: clearance of rales/ crackles, decrease in JVD, reduction in peripheral edema, decrease in BNP by at least 20%, no evidence of pulmonary edema on CXR.

Exclusion Criteria: ACUTE HEART FAILURE

1. NYHA class III/ IV despite treatment with diuretics.
2. Co-existent pulmonary disease such as asthma/ COPD/ interstitial lung disease.
3. Known allergy to electrode gel and medical adhesive used on electrocardiographic electrodes.
4. Pregnancy (as any effect of this device use on pregnancy is not known)..
5. Patient belonging to a vulnerable population such as institutionalized persons, prisoners and persons with decisional incapacity or dementia.
6. Presence of severe aortic regurgitation.
7. Second degree Mobitz type II or third degree heart block, unless treated with a cardiac pacemaker.
8. Implantation of a left ventricular assist device, hemodynamic monitor, activated minute ventilation pacemaker, or biventricular pacemaker (Cardiac Resynchronization Therapy) with the V-to-V interval set at more than 5 milliseconds offset.
9. Implantation of a cardiac resynchronization device within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the changes in cardiac hemodynamic parameters (Cardiac output, cardiac index, and thoracic fluid content) between normal, acute HF and chronic HF subjects with a trial of controlled slow breathing with biofeedback. | Half hour

CONTACTS AND LOCATIONS:
Overall Officials: Darshak H Karia, MD, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Albert Einstein Healthcare Network, Philadelphia, Pennsylvania, United States